CLINICAL TRIAL: NCT03371706
Title: Communication Bridge: A Person-centered Internet-based Intervention for Individuals With Primary Progressive Aphasia
Brief Title: Communication Bridge 2
Acronym: CB2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB23-1334; 1R01AG055425-01A1 (NIH)
Record Dates: First submitted 2017-12-08; First posted 2017-12-13 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-08

CONDITIONS: Primary Progressive Aphasia
Keywords: aphasia; primary progressive aphasia; dementia; communication; frontotemporal dementia; Alzheimer's disease
MeSH Terms: conditions — Aphasia, Primary Progressive; Aphasia; Dementia; Communication; Frontotemporal Dementia; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: NIH Stage 2 behavioral clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Communication Bridge™ (Experimental): Participants receive Communication Bridge™, a multi-component, participation-focused, dyadic intervention in which both the person with PPA and their co-enrolled communication partner are intervention recipients. Communication Bridge™ is modelled on the Living with Aphasia: Framework for Outcome Measurement (A-FROM) and the Care Pathway Model that was developed for persons living with primary progressive aphasia. Consistent with participation-focused intervention models personally salient training stimuli are incorporated into all therapy activities in the Experimental arm.
  Interventions: Behavioral: Communication Bridge™
- Evidence-Based Impairment Focused (Active Comparator): The Control arm includes a non-dyadic intervention in which the person with PPA is the active intervention recipient and their communication partner is in a supporting role. In the Control arm, participants receive a speech-language intervention designed to address impairment and functional limitations, comprised of activities that address word retrieval and 'automatic' speech production using fixed, non-personalized, stimuli across participants.
  Interventions: Behavioral: Evidence-Based Impairment Focused

INTERVENTIONS:
Behavioral: Communication Bridge™ — Evidence-based speech language therapy treatment will be compared and contrasted in the two arms of the study.
  Arms: Communication Bridge™
Behavioral: Evidence-Based Impairment Focused — Evidence-based speech language therapy treatment will be compared and contrasted in the two arms of the study.
  Arms: Evidence-Based Impairment Focused

SUMMARY:
This study will use a randomized controlled trial design to evaluate the effect of two evidence-based treatments for adults with mild Primary Progressive Aphasia (PPA). The aim of the study is to help us better understand the effects of speech language therapy on communication abilities in individuals with PPA.

Participants with a diagnosis of PPA and their actively-engaged care partners will be involved in the study for 12 months. Each participant will receive a laptop equipped with the necessary applications and features for the study. Participants will receive 5 evaluations and 15 speech therapy sessions with a licensed speech therapist, as well as access to Communication Bridge, a personalized web application to practice home exercises that reinforce treatment strategies. There are no costs to participate in this study.

ELIGIBILITY:
Inclusion Criteria (person with PPA):

1. Meets diagnostic criteria for PPA based on neurologist and supporting medical assessments (extracted from medical records)
2. English as primary language used in daily communication activities (by self-report)
3. Adequate hearing (aided or unaided) for communicating with others in a crowded room (by self-report)
4. Adequate vision (aided or unaided) for reading a newspaper, or other functional materials (by self-report)
5. Able to pass technology screening and demonstrates sufficient knowledge for use of video conference and Communication Bridge™ web application use (with or without training)
6. Geriatric Depression Scale score ≤ 9
7. Mild-moderate PPA informed by a structured interview with a speech-language pathologist and a standardized testing battery.

Inclusion Criteria (Co-enrolled communication partner):

1. 18+ years of age
2. English as primary language used in daily communication activities (by self-report)
3. Adequate hearing (aided or unaided) for communicating with others in a crowded room (by self-report)
4. Able to pass technology screening* and demonstrates sufficient knowledge for use of video conference and Communication Bridge™ web application use (with or without training)

Exclusion Criteria:

* A dementia diagnosis other than Primary Progressive Aphasia
* Participation is co-enrolled in an outside speech language therapy program during the study course.
* Communication partners will be excluded if they have a pre-existing communication impairment that would affect study participation (e.g., aphasia, dementia)

Medical records will be requested and reviewed to determine eligibility.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Rogalski, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- The Healthy Aging & Alzheimer's Research Care Center (University of Chicago), Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Publication of study protocol manuscript prior to enrolling final participant. Communication Bridge Manual of Procedures upon publication of study protocol or when final participant completes all study procedures (whichever comes later). Statistical Analysis Plan to be published with study protocol.
Access Criteria: With approval of study administration team, with the exception of documents that will be made available to the public following study completion (manual of procedures). Analyzed and processed data will be available by request with an approved Collaborator Agreement.

REFERENCES:
- [Derived] Roberts AC, Rademaker AW, Salley EA, Mooney A, Morhardt D, Fried-Oken M, Weintraub S, Mesulam M, Rogalski E. Communication Bridge-2 (CB2): an NIH Stage 2 randomized control trial of a speech-language intervention for communication impairments in individuals with mild to moderate primary progressive aphasia. Trials. 2022 Jun 13;23(1):487. doi: 10.1186/s13063-022-06162-7. PMID 35698099
- [Derived] Mesulam MM, Coventry C, Kuang A, Bigio EH, Mao Q, Flanagan ME, Gefen T, Sridhar J, Geula C, Zhang H, Weintraub S, Rogalski EJ. Memory Resilience in Alzheimer Disease With Primary Progressive Aphasia. Neurology. 2021 Feb 9;96(6):e916-e925. doi: 10.1212/WNL.0000000000011397. Epub 2021 Jan 13. PMID 33441454

RESULTS

PARTICIPANT FLOW:
Groups:
- Communication Bridge™ (Persons With Primary Progressive Aphasia); Communication Bridge™ (Care Partners: Participants receive Communication Bridge™, a multi-component, participation-focused, dyadic intervention in which both the person with PPA and their co-enrolled communication partner are intervention recipients. Communication Bridge™ is modelled on the Living with Aphasia: Framework for Outcome Measurement (A-FROM) and the Care Pathway Model that was developed for persons living with primary progressive aphasia. Consistent with participation-focused intervention models personally salient training stimuli are incorporated into all therapy activities in the Experimental arm.
  Communication Bridge™: Evidence-based speech language therapy treatment will be compared and contrasted in the two arms of the study.
- Evidence-Based Impairment Focused (Persons With Primary Progressive Aphasia); Evidence-Based Impairment Focused (Care Partners): The Control arm includes a non-dyadic intervention in which the person with PPA is the active intervention recipient and their communication partner is in a supporting role. In the Control arm, participants receive a speech-language intervention designed to address impairment and functional limitations, comprised of activities that address word retrieval and 'automatic' speech production using fixed, non-personalized, stimuli across participants.
  Evidence-Based Impairment Focused: Evidence-based speech language therapy treatment will be compared and contrasted in the two arms of the study.
Period: Overall Study
Arm/Group | Communication Bridge™ (Persons With Primary Progressive Aphasia) | Communication Bridge™ (Care Partners | Evidence-Based Impairment Focused (Persons With Primary Progressive Aphasia) | Evidence-Based Impairment Focused (Care Partners)
Started | 56 | 56 | 39 | 39
Completed | 50 | 50 | 39 | 39
Not Completed | 6 | 6 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Communication Bridge™ (Persons With Primary Progressive Aphasia) | Evidence-Based Impairment Focused (Persons With Primary Progressive Aphasia) | Total
Number analyzed (Participants) | 56 | 39 | 95
Age, Customized [Mean (Standard Deviation); unit: years]
  Age at baseline | 66.9 (7.2) | 67.4 (7.8) | 67.1 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 49
  Male | 31 | 15 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 56 | 38 | 94
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 56 | 37 | 93
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Years of education [Mean (Standard Deviation); unit: years] | 16.2 (2.5) | 16.7 (2.3) | 16.4 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Communication Confidence (CCRSA)
Description: Communication Confidence Rating Scale in Aphasia, a 0-100 numeric rating scale with 0 representing 'not confident' and 100 representing 'very confident'. Higher scores indicate greater confidence.
Time Frame: 5 assessment time points through study completion - Baseline, Post Intervention 1 (3 months), Six months, Post Intervention 2 (9 months), and 12 months
Population: the number analyzed in some rows differs from the overall number analyzed due to participant withdrawal and missing data.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Communication Bridge™ (Person With Primary Progressive Aphasia): Participants receive Communication Bridge™, a multi-component, participation-focused, dyadic intervention in which both the person with PPA and their co-enrolled communication partner are intervention recipients. Communication Bridge™ is modelled on the Living with Aphasia: Framework for Outcome Measurement (A-FROM) and the Care Pathway Model that was developed for persons living with primary progressive aphasia. Consistent with participation-focused intervention models personally salient training stimuli are incorporated into all therapy activities in the Experimental arm.
  Communication Bridge™: Evidence-based speech language therapy treatment will be compared and contrasted in the two arms of the study.
- Evidence-Based Impairment Focused (Person With Primary Progressive Aphasia): The Control arm includes a non-dyadic intervention in which the person with PPA is the active intervention recipient and their communication partner is in a supporting role. In the Control arm, participants receive a speech-language intervention designed to address impairment and functional limitations, comprised of activities that address word retrieval and 'automatic' speech production using fixed, non-personalized, stimuli across participants.
  Evidence-Based Impairment Focused: Evidence-based speech language therapy treatment will be compared and contrasted in the two arms of the study.
Arm/Group | Communication Bridge™ (Person With Primary Progressive Aphasia) | Evidence-Based Impairment Focused (Person With Primary Progressive Aphasia)
Number analyzed (Participants) | 56 | 39
units on a scale
  Baseline | 72.6 (1.8) | 72.9 (2.6)
  Post Intervention 1 (3 months): number analyzed (Participants) | 53 | 39
  Post Intervention 1 (3 months) | 73.7 (1.9) | 74.5 (2.4)
  Six Months: number analyzed (Participants) | 51 | 39
  Six Months | 72.1 (2.1) | 73.1 (2.5)
  Post Intervention 2 (9 months): number analyzed (Participants) | 50 | 39
  Post Intervention 2 (9 months) | 72.2 (2.2) | 71.6 (2.5)
  12 Months: number analyzed (Participants) | 50 | 37
  12 Months | 69.1 (2.7) | 70.1 (2.5)

2. Primary Outcome: Change in Communication Participation Item Bank (CPIB)
Description: Communication Participation Item Bank is a 4-point rating scale with 0 representing 'very much' and 3 representing 'not at all'. Higher scores indicate greater severity of communication challenges.
  We are reporting on change in CPIB scores using T-scores. The Communicative Participation Item Bank (CPIB) T-score range is as follows:
  T57.5 and above: Represents a "normal" experience of communicative participation or "minimal problems" T57.5-T45: Represents mild challenges T45-T35: Represents moderate challenges T35 and below: Represents severe challenges
  The CPIB is a patient-reported instrument that measures communicative participation. The mean T-score is 50, and the standard deviation is 10. Higher scores are more favorable, indicating less interference in participation. The ideal score, or someone who reports no problems with communicative participation, would be a T-score of 74.3
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Communication Bridge™ (Person With Primary Progressive Aphasia) | Evidence-Based Impairment Focused (Person With Primary Progressive Aphasia)
Number analyzed (Participants) | 56 | 39
units on a scale
  Baseline | 46.0 (0.8) | 47.1 (1.0)
  Post Intervention 1 (3 months): number analyzed (Participants) | 53 | 39
  Post Intervention 1 (3 months) | 47.4 (0.9) | 47.7 (1.9)
  Six Months: number analyzed (Participants) | 52 | 39
  Six Months | 45.6 (1.0) | 46.8 (1.1)
  Post Intervention 2 (9 months): number analyzed (Participants) | 50 | 39
  Post Intervention 2 (9 months) | 46.0 (0.9) | 46.3 (1.0)
  12 Months: number analyzed (Participants) | 50 | 38
  12 Months | 45.5 (1.0) | 45.0 (1.0)

3. Primary Outcome: Change in Communication Participation Person Centered Goals
Description: This measure assesses progress toward communication participation goals using Goal Attainment Scaling (GAS). Participants developed personalized goals, each set to a baseline value of '0'. Progress was tracked using a 7-point scale, where -3 represents 'no longer participating' and +3 represents 'exceeded goal'. Higher scores indicate better progress toward goal achievement. Goals were evaluated at 3, 6, 9, and 12 months, with the results reported as the percentage of goals that:
  Worsened (scores of -1, -2, or -3) No change (score remained at 0) Improved (scores of +1, +2, or +3), including getting close to, reaching, or exceeding the goal.
  The table below presents the percentage of goals falling into each of these categories at each assessment point.
Time Frame: 4 assessment time points through study completion - Post Intervention 1 (3 months), Six months, Post Intervention 2 (9 months), and 12 months
Measure: Number; unit: percentage of goals
Units Other Than Participants: Number of Goals
Arm/Group | Communication Bridge™ (Person With Primary Progressive Aphasia) | Evidence-Based Impairment Focused (Person With Primary Progressive Aphasia)
Number analyzed (Participants) | 53 | 39
Number analyzed (Number of Goals) | 159 | 116
percentage of goals
  Post Intervention 1 - (Worse than baseline) | 3.8 | 6.9
  Post Intervention 1 - (No change from baseline) | 29.6 | 44.0
  Post Intervention 1 - (Getting close to, reached, or exceed) goal | 66.7 | 49.1
  Six Months - (Worse than baseline) | 16.3 | 18.0
  Six Months - (No change from baseline) | 23.5 | 35.0
  Six Months - (Getting close to , reached, or exceeded expected goal) | 60.1 | 47.0
  Post Intervention 2 - (Worse than baseline) | 16.0 | 18.8
  Post Intervention 2 - (No change from baseline) | 22.0 | 26.5
  Post Intervention 2 - (Getting close to, reached or exceeded expected goal) | 62.0 | 54.7
  12 Months (Worse than baseline) | 21.3 | 20.2
  12 Months - (No change from baseline) | 18.0 | 23.7
  12 Months - (Getting close to, reached or exceeded expected goal) | 60.7 | 56.1

4. Other Pre Specified Outcome: Change in Word Accuracy (Trained Words)
Description: proportion of participants accuracy on trained words. Higher values indicate greater number of words produced after first prompt. Range 0 - 30
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: words
Arm/Group | Communication Bridge™ (Person With Primary Progressive Aphasia) | Evidence-Based Impairment Focused (Person With Primary Progressive Aphasia)
Number analyzed (Participants) | 56 | 39
words
  Baseline | 18.2 (1.0) | 13.6 (1.1)
  Post Intervention 1 (PIE1) (3 months) | 25.2 (0.8) | 25.1 (1.0)
  Six Months | 23.6 (1.0) | 23.5 (1.0)
  Post Intervention 2 (PIE2) (9 months) | 25.1 (0.9) | 23.7 (1.1)
  12 months | 22.7 (1.1) | 21.8 (1.2)

5. Other Pre Specified Outcome: Change in Script Accuracy (Trained Scripts)
Description: proportion of participants accuracy on trained scripts. Higher values indicate greater level of script performance as a proportion. Range 0 - 1.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: proportion of accuracy
Arm/Group | Communication Bridge™ (Person With Primary Progressive Aphasia) | Evidence-Based Impairment Focused (Person With Primary Progressive Aphasia)
Number analyzed (Participants) | 56 | 39
proportion of accuracy
  Baseline | 0.23 (0.03) | 0.27 (0.03)
  Post Intervention 1 (PIE1) (3 months) | 0.59 (0.05) | 0.64 (0.06)
  Six Months | 0.60 (0.05) | 0.62 (0.06)
  Post Intervention 2 (PIE2) (9 months) | 0.66 (0.04) | 0.70 (0.05)
  12 Months | 0.60 (0.05) | 0.55 (0.06)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Communication Bridge™ | Evidence-Based Impairment Focused
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/39
Serious Adverse Events (participants affected / at risk) | 7/56 | 4/39
Other Adverse Events (participants affected / at risk) | 5/56 | 7/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Communication Bridge™ (N=56) | Evidence-Based Impairment Focused (N=39)
Medical event (Surgical and medical procedures) | 6 (6) | 4 (6)
Psychosocial events (Social circumstances) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Communication Bridge™ (N=56) | Evidence-Based Impairment Focused (N=39)
Frustration/Fatigue due to cognitive testing (Social circumstances) | 1 (1) | 0 (0)
Frustration/Fatigue due to therapy sessions (Social circumstances) | 1 (1) | 0 (0)
Psychosocial events (Social circumstances) | 3 (3) | 7 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT03371706/Prot_SAP_000.pdf